CLINICAL TRIAL: NCT01998984
Title: Efficacy and Safety of Ingenol Mebutate Gel 0.06% When Applied Once Daily for 2, 3 or 4 Consecutive Days to a Treatment Area of Approximately 250 cm2 on Trunk and Extremities in Subjects With Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0105-1020
Record Dates: First submitted 2013-11-21; First posted 2013-12-03 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2018-11

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2 days placebo and 2 days drug (Experimental): Placebo and drug
  Interventions: Drug: ingenol mebutate; Other: Placebo
- 1 day placebo and 3 days drug (Experimental): Placebo and drug
  Interventions: Drug: ingenol mebutate; Other: Placebo
- 4 days placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 4 days drug (Experimental): Drug
  Interventions: Drug: ingenol mebutate

INTERVENTIONS:
Drug: ingenol mebutate
  Arms: 1 day placebo and 3 days drug; 2 days placebo and 2 days drug; 4 days drug
Other: Placebo
  Arms: 1 day placebo and 3 days drug; 2 days placebo and 2 days drug; 4 days placebo

SUMMARY:
This is a randomised, double-blind, parallel groups, vehicle controlled, 8-week phase 2 trial. The objective is to evaluate efficacy of ingenol mebutate gel 0.06 % after once daily treatment for 2, 3 or 4 consecutive days compared to vehicle gel

ELIGIBILITY:
Inclusion Criteria:

Subjects with 5 to 20 clinically typical, visible and discrete AKs within a contiguous area of approximately 250 cm² sun-damaged skin on either trunk (except chest), or extremities

Exclusion Criteria:

* Location of the treatment area (trunk (except chest) or extremities)

  * within 5 cm of an incompletely healed wound,
  * within 5 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC)
* Prior treatment with ingenol mebutate within the selected treatment area
* Lesions in the treatment area that have:

  * atypical clinical appearance (e.g., hypertrophic,hyperkeratotic or cutaneous horns) and/or,
  * recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Siegel, MD, MS, Principal Investigator — Lond Island Skin Cancer and Dermatologic Surgery
Locations (1):
- Long Island Skin Cancer and Dermatologic Surgery, Smithtown, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were followed for 8 weeks following the first application of investigational medicinal product (IMP) at Day 1 (4-day treatment period including an 8-week follow-up period).
Pre-assignment Details: 266 participants were enrolled of which 224 participants were randomized to treatment
Groups:
- Ingenol 2 Days: Ingenol mebutate gel 0.06% and vehicle gel applied topically once daily to a contiguous area of approximately 250 cm2 sun-damaged skin on trunk (except chest), or extremities (arm with or without back of hand, or leg). Vehicle gel was applied for 2 days and ingenol mebutate gel 0.06% was applied for 2 days for a total 4 consecutive days.
- Ingenol 3 Days: Ingenol mebutate gel 0.06% and vehicle gel applied topically once daily to a contiguous area of approximately 250 cm2 sun-damaged skin on trunk (except chest), or extremities (arm with or without back of hand, or leg). Vehicle gel was applied for 1 day and ingenol mebutate gel 0.06% was applied for 3 days for a total 4 consecutive days.
- Ingenol 4 Days: Ingenol mebutate gel 0.06% applied topically once daily to a contiguous area of approximately 250 cm2 sun-damaged skin on trunk (except chest), or extremities (arm with or without back of hand, or leg) for 4 consecutive days.
- Vehicle: Vehicle gel applied topically once daily to a contiguous area of approximately 250 cm2 sun-damaged skin on trunk (except chest), or extremities (arm with or without back of hand, or leg) for 4 consecutive days.
Period: Overall Study
Arm/Group | Ingenol 2 Days | Ingenol 3 Days | Ingenol 4 Days | Vehicle
Started | 55 | 59 | 49 | 61
Completed | 55 | 58 | 48 | 58
Not Completed | 0 | 1 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ingenol 2 Days: 2 days treatment with ingenol mebutate 0.06% gel and 2 days treatment with vehicle gel
- Ingenol 3 Days: 3 days treatment with ingenol mebutate 0.06% gel and 1 day treatment with vehicle gel
- Ingenol 4 Days: 4 days treatment with ingenol mebutate 0.06% gel
- Vehicle: 4 days treatment with vehicle gel
- Total: Total of all reporting groups
Arm/Group | Ingenol 2 Days | Ingenol 3 Days | Ingenol 4 Days | Vehicle | Total
Number analyzed (Participants) | 55 | 59 | 49 | 61 | 224
Age, Continuous [Mean (Full Range); unit: years] | 67.7 [39 to 88] | 68.1 [42 to 87] | 68.8 [44 to 89] | 68.6 [42 to 91] | 68.3 [39 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 27 | 13 | 20 | 80
  Male | 35 | 32 | 36 | 41 | 144
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 26 | 17 | 25 | 92
  Australia | 31 | 33 | 32 | 36 | 132

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Clearance of Actinic Keratosis Lesions (AKs)
Description: Complete clearance of AKs at Week 8 was defined as a 100% reduction from baseline in number of AKs.
  The table presents the mean across 1000 multiple imputations. Missing values for AK count were imputed sequentially from a negative binomial regression model with treatment group, AK counts at the previous visit, and analysis site as covariates and log baseline AK count as offset.
Time Frame: At Week 8
Population: The analysis was based on the Full Analysis Set, which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Ingenol 3 Days: 1 day treatment with vehicle gel and 3 days treatment with ingenol mebutate 0.06% gel
Arm/Group | Ingenol 2 Days | Ingenol 3 Days | Ingenol 4 Days | Vehicle
Number analyzed (Participants) | 55 | 59 | 49 | 61
percentage of participants | 12.7 | 5.1 | 26.8 | 0.0
Statistical Analysis 1: Comparison: Ingenol 3 Days vs Vehicle; Treatment comparison based on 1000 imputations of AK count at week 8 using a negative binomial regression model with factors treatment and analysis site and with log of baseline AK count as offset. Cochran-Mantel-Haenszel logit estimators were used for comparisons with vehicle due to absence of cleared participant in the vehicle group; Test type: Superiority; p = 0.18, Cochran-Mantel-Haenszel — P-value was adjusted for analysis site using Rubin's pooling methodology after log transformation of RR (relative risk) of each imputation. Complete clearance relative to vehicle group and 2-day group; Relative risk = 2.97, 95% CI 2-sided [0.60 to 14.74] — Relative risk and confidence interval were adjusted for analysis site using Rubin's pooling methodology after log transformation of RR of each imputation. Complete clearance relative to vehicle group and 2-day group
Statistical Analysis 2: Comparison: Ingenol 2 Days vs Vehicle; Treatment comparison based on 1000 imputations of AK count at week 8 using a negative binomial regression model with factors treatment and analysis site and with log of baseline AK count as offset. Cochran-Mantel-Haenszel logit estimators were used for comparisons with vehicle due to absence of cleared subject in the vehicle group. Type I error not controlled; Test type: Superiority; p = 0.051, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Relative risk = 3.51, 95% CI 2-sided [1.00 to 12.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Ingenol 2 Days vs Ingenol 3 Days; Treatment comparison based on 1000 imputations of AK count at week 8 using a negative binomial regression model with factors treatment and analysis site and with log of baseline AK count as offset. Type I error not controlled. Mantel-Haenszel estimators were used; Test type: Superiority; p = 0.25, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Relative risk = 0.47, 95% CI 2-sided [0.13 to 1.68] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Reduction in Actinic Keratosis (AK) Lesion Count From Baseline (Day 1) (Multiple Imputation)
Description: The number of clinically visible AK lesions identified in the treatment area was to be recorded at Visit 1(≤14 days prior to Day 1).
  The analysis was based on 1000 imputations of actinic keratosis lesion count at Week 8 using a negative binomial regression model with factors treatment and analysis site and with log of baseline actinic keratosis lesion count as offset. The table shows the adjusted percentage reduction from baseline.
  Values for the Ingenol 4 days arm were calculated separately based on observed cases. On the basis of the data monitoring committee's recommendation the 4-day active treatment group was closed, and this arm was excluded from statistical models and comparisons in the secondary efficacy analyses.
Time Frame: At Week 8
Population: The analysis was based on the Full Analysis Set, which was defined as all randomized participants.
Measure: Mean (95% Confidence Interval); unit: percentage of reduction
Arm/Group | Ingenol 2 Days | Ingenol 3 Days | Ingenol 4 Days | Vehicle
Number analyzed (Participants) | 55 | 59 | 48 | 61
percentage of reduction | 64.5 [57.8 to 70.2] | 68.3 [62.4 to 73.4] | 73.6 [65.8 to 81.5] | 11.9 [-2.2 to 24.1]
Statistical Analysis 1: Comparison: Ingenol 2 Days vs Vehicle; Test type: Superiority; p < 0.001, Negative binomial regression — P-value was from negative binomial regression model with factors treatment and analysis site and with log of baseline AK count as offset with 1000 Imputations; Ratio of adjusted mean = 0.40, 95% CI 2-sided [0.32 to 0.51] — Estimation parameter and confidence interval were from negative binomial regression model with factors treatment and analysis site and with log of baseline AK count as offset with 1000 Imputations
Statistical Analysis 2: Comparison: Ingenol 3 Days vs Vehicle; Test type: Superiority; p < 0.001, Negative binomial regression — [p-value comment as in outcome 2, analysis 1]; Ratio of adjusted mean = 0.36, 95% CI 2-sided [0.29 to 0.45] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Ingenol 2 Days vs Ingenol 3 Days; Test type: Superiority; p = 0.36, Negative binomial regression — [p-value comment as in outcome 2, analysis 1]; Ratio of adjusted mean = 0.89, 95% CI 2-sided [0.70 to 1.14] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With Partial Clearance of AKs
Description: Partial clearance of AKs at Week 8, defined as at least 75% reduction from baseline in number of AKs, was analysed in the same way as the primary response criterion.
  The percent reduction at Week 8 from baseline was analyzed using a negative binomial regression for the AK count at Week 8 with treatment group and pooled sites as factors and baseline count as offset variable (using multiple imputations to account for missing values).
  The table presents the mean across 1000 multiple imputations. Missing values for AK count were imputed sequentially from a negative binomial regression model with treatment group, AK counts at the previous visit, and analysis site as covariates and log baseline AK count as offset.
Time Frame: At Week 8
Population: The analysis was based on the Full Analysis Set, which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Ingenol 2 Days | Ingenol 3 Days | Ingenol 4 Days | Vehicle
Number analyzed (Participants) | 55 | 59 | 49 | 61
percentage of participants | 47.3 | 56.2 | 60.4 | 2.0
Statistical Analysis 1: Comparison: Ingenol 3 Days vs Vehicle; The treatment comparison was based on 1000 imputations of AK count at week 8 using a negative binomial regression model with factors treatment and analysis site and with log of baseline AK count as offset; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P value adjusted for analysis site; Relative risk = 32.26, 95% CI 2-sided [4.39 to 236.8] — Relative risk and confidence interval were adjusted for analysis site and were Mantel-Haenszel estimators. Relative risk of partial clearance relative to vehicle group
Statistical Analysis 2: Comparison: Ingenol 2 Days vs Vehicle; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — Adjusted for analysis site. Relative risk of partial clearance relative to vehicle group; Relative risk = 25.20, 95% CI 2-sided [3.39 to 187.4] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Ingenol 2 Days vs Ingenol 3 Days; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.28, Cochran-Mantel-Haenszel — Adjusted for analysis site. Relative risk of partial clearance relative to 2-day group; Relative risk = 1.20, 95% CI 2-sided [0.86 to 1.65] — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: From Day 1 to Week 8 (Day 56)
Arm/Group | Ingenol 2 Days | Ingenol 3 Days | Ingenol 4 Days | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/59 | 0/49 | 0/61
Serious Adverse Events (participants affected / at risk) | 3/55 | 5/59 | 4/49 | 0/61
Other Adverse Events (participants affected / at risk) | 48/55 | 55/59 | 47/49 | 7/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol 2 Days (N=55) | Ingenol 3 Days (N=59) | Ingenol 4 Days (N=49) | Vehicle (N=61)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 3 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol 2 Days (N=55) | Ingenol 3 Days (N=59) | Ingenol 4 Days (N=49) | Vehicle (N=61)
Application site pain (General disorders) | 45 | 50 | 43 | 3
Application site pruritus (General disorders) | 19 | 27 | 14 | 2
Application site discomfort (General disorders) | 2 | 3 | 2 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting or presenting a manuscript relating to the clinical trial to a publisher, reviewer or other outside person, the investigator shall provide to LEO Pharma A/S a copy of all such manuscripts, and LEO Pharma A/S shall have rights to review and comment. Upon the request of LEO Pharma A/S the investigator shall remove any confidential information (other than results generated by the investigator) prior to submitting or presenting the manuscripts.